CLINICAL TRIAL: NCT01042106
Title: A Randomized, Double-blind, Placebo-controlled, Multiple Ascending Oral Dose Study to Evaulate Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of DSP-8658 in Type 2 Diabetic and Healthy Subjects
Brief Title: Safety, Pharmacokinetics and Pharmacodynamics of DSP-8658 in Patients With Type 2 Diabetes Mellitus and Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D6950153
Record Dates: First submitted 2009-12-21; First posted 2010-01-05 (Estimated); Last update posted 2013-09-16 (Estimated); Status verified 2013-09

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- DSP-8658 (Experimental): DSP-8658 2.5, 10, 20, 40 mg once daily
  Interventions: Drug: DSP-8658
- Placebo (Placebo Comparator): Placebo 2.5, 10, 20, and 40 mg doses once daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: DSP-8658 — Ascending doses of DSP-8658 - 2.5, 10, 20, 40 mg orally once daily
  Arms: DSP-8658
Drug: Placebo — Placebo 2.5, 10, 20, 40 mg orally once daily
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics of multiple ascending doses of DSP-8658 in patients with Type 2 diabetes mellitus and healthy adults.

ELIGIBILITY:
Inclusion Criteria: Diabetic subjects

* Age ≥ 18 and ≤ 65 years
* Body Mass Index ≤45
* Drug naive type 2 diabetes or type 2 diabetes previously treated with an oral antidiabetic drug

Inclusion Criteria: Healthy subjects

* Age ≥ 18 and ≤ 65 years
* Body Mass Index ≥ 18 and ≤ 29
* Good health as determined by medical history, ECG, clinical chemistry, hematology, urinalysis, virology, and a physical examination.

Exclusion Criteria: Diabetic subjects

* Have a current or expected requirement for any antidiabetic or lipid-lowering drug

Exclusion Criteria: Healthy subjects

* Have, or have had a history of clinically significant neurological, urological, gastrointestinal, renal, hepatic, cardiovascular, psychological, pulmonary, metabolic, endocrine, hematological, or other major disorders including cancer

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-11; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Safety assessments include physical examination, laboratory variables and ECG. | 20 days

SECONDARY OUTCOMES:
Pharmacokinetics of DSP-8658 and its metabolites: levels of DSP-8658 and its metabolites will be measured and analyzed at various time points throughout the study. | 20 days
Pharmacodynamics of DSP-8658 (how DSP-8658 acts in the body to affect glucose and lipid control): glucose and lipid levels will be measured at various time points throughout the study. | 18 days

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, MD, Study Director — Sumitomo Pharma America, Inc.
Locations (1):
- Cetero Research, San Antonio, Texas, United States